CLINICAL TRIAL: NCT02060331
Title: Severe Pelvic Organ Prolapse and Post-Obstructive Diuresis (SOPPO) Pilot Study
Acronym: SOPPO
Status: Withdrawn | Type: Observational
Why Stopped: Difficult to recruit to.
Sponsor: Loyola University (Other)
Responsible Party: Principal Investigator, Elizabeth Mueller, Principal Investigator, Loyola University
Other Study IDs: 206058
Record Dates: First submitted 2014-02-10; First posted 2014-02-12 (Estimated); Last update posted 2016-06-02 (Estimated); Status verified 2016-06

CONDITIONS: Nocturia; Pelvic Organ Prolapse
Keywords: Nocturia; Pelvic Organ Prolapse; Nocturnal Polyuria; Post-obstructive Diuresis
MeSH Terms: conditions — Nocturia; Pelvic Organ Prolapse

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — The awake and asleep renal nocturia urine panels will require the patient to collect her urine output into two laboratory provided basins for one twenty-four hour period. The "renal nocturia, awake" urine panel will be obtained from urine collected from 0600-1800. The "renal nocturia, asleep" urine panel will be obtained from urine collected from 1800-0600, ie through the following day.
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Pelvic Organ Prolapse with Nocturia: Pelvic Organ Prolapse with Nocturia

SUMMARY:
In our experience, women with severe pelvic organ prolapse (POP) frequently have bothersome nocturia. The International Continence Society (ICS) defines nocturia as "having to wake at night one or more times to void." Though some of this nocturia may be secondary to obstructed bladder emptying, the investigators hypothesize that in some women compression of the bilateral ureters due to prolapsed pelvic organs during the day and subsequent relief of that prolapse while the patient lays supine overnight results in nighttime post-obstructive diuresis (inability to concentrate urine) and resultant large nighttime urine volumes and nocturia. Previous case reports have proposed that vaginal and uterine vault prolapse causes obstruction due to descent of the bladder floor which leads to compression of the bilateral ureters between the uterus and the borders of the genital opening. No large prospective studies, however, have evaluated the possible impact of this phenomenon on patients or the possible post-operative changes following surgical correction of POP.

Using the Nocturnal Enuresis, and Sleep interruption Questionnaire (NNES-Q), voiding diaries, and urine studies, the investigators aim to evaluate the pre-operative and post-operative voiding habits and urinary parameters of women with severe pelvic organ prolapse and bothersome nocturia who undergo colpocleisis. Colpocleisis is a procedure which surgically obliterates the vaginal lumen to treat severe POP in properly counseled patients with >90% satisfaction rates. Other treatments offered to women, such as the laparoscopic or open sacrocolpopexy, uterosacral ligament suspension, and sacrospinous ligament suspension, also offer high rates of success. The investigators aim to determine whether surgical correction of severe pelvic organ prolapse, to be defined as either with colpocleisis, laparoscopic or open sacrocolpopexy, uterosacral ligament suspension, or sacrospinous ligament suspension, results in improvement and/or resolution of nocturia and post-obstructive diuresis.

DETAILED DESCRIPTION:
1. Significance or Clinical Relevance of Project:

   Numerous women undergo pelvic organ prolapse surgery every year. The most common reasons for surgical management of POP include symptoms immediately related to the prolapsing organs, such as pelvic pressure, vaginal bulge sensation, vaginal mucosal irritation, as well as defecatory dysfunction, limitations on sexual intercourse, and aesthetic dissatisfaction. When counseling patients about possible surgical management of POP, clinicians would be remiss if they did not address the potential quality of life improvement surgery may provide from a urinary standpoint, as well as possible decreased risk of renal failure. Stress and urge incontinence and urinary urgency are frequently alleviated by restoration of the pelvic floor support, however, nocturia may be treated as well.
2. Relevant Research of Others:

   Several case reports exist describing urinary obstruction, bilateral hydronephrosis, and acute or chronic renal failure that can occur with severe pelvic organ prolapse. No larger scale prospective descriptive studies exist, however, demonstrating the urinary symptoms or pathophysiology behind the urinary tract obstruction that may accompany pelvic organ prolapse. Also, no prospective studies exist to evaluate the improvement in those symptoms and relief of physiologic obstruction after surgical correction of pelvic organ prolapse.
3. Methods/Materials:

Women referred to the urogynecology clinic for management of apical Stage III-IV POP with bothersome nocturia as noted in their initial urogynecologic evaluation who opt for surgical management will be identified for inclusion in the study. In addition to routine urogynecologic and pre-operative work-up, after consenting for the study, they will be asked to complete pre- and post-operative Nocturia, Nocturnal Enuresis, and Sleep interruption Questionnaires (NNES-Q) (appendix), voiding diaries (appendix), and awake and asleep renal nocturia urine panels. Women will serve as their own pre- and post-operative control subjects.

Enrolled patients will be educated on how to perform the voiding diary and awake and asleep renal nocturia urine panel. The voiding diary will require the patient to measure the date, time, voided urine amount (using a urine hat placed over a toilet), degree of incontinence (dry, moist, soaked), presence or absence of urge to urinate, activity immediately prior to urination episode, and fluid intake for three non-consecutive twenty-four hour periods. The awake and asleep renal nocturia urine panels will require the patient to collect her urine output into two laboratory provided basins for one twenty-four hour period. The "renal nocturia, awake" urine panel will be obtained from urine collected from 0600-1800. The "renal nocturia, asleep" urine panel will be obtained from urine collected from 1800-0600, ie through the following day.

Six to thirteen weeks post-operatively, enrolled patients will be asked to repeat the NNES-Q questionnaire, voiding diary, and awake and asleep renal nocturia urine panels as described above.

Patients who complete all of the aforementioned questionnaires and studies will be reimbursed with a $25 check. This compensation will be disclosed to potential study candidates prior to enrollment in the study.

The data obtained will be de-identified and then entered into SPSS v. 20 software for statistical analysis.

ELIGIBILITY:
Inclusion Criteria:

* Female gender
* Bothersome nocturia (presence of ≥1 void per night averaged over 4 weeks with ≥5/10 on 0-10 bother scale)
* Age >18 years
* Apical stage III-IV pelvic organ prolapse as defined by the Pelvic Organ Prolapse Quantification (POP-Q) Staging Criteria: Stage III - leading edge > +1 cm but < +(total vaginal length-2) cm, Stage IV - leading edge ≥ +(tvl-2) cm
* Undergoing surgical correction (colpocleisis, laparoscopic or open sacrocolpopexy, uterosacral ligament suspension, or sacrospinous ligament suspension) for POP by Drs. Mueller, Brincat, and/or Brubaker

Exclusion Criteria:

* Obstructive sleep apnea (clinically diagnosed on sleep study or patients with excessive daytime sleepiness or nighttime apneic periods as identified by patient or spouse)
* Diuretic use (ie for hypertension)
* Renal insufficiency (Chronic Kidney Disease Stage 3-5, measured or estimated Glomerular Filtration Rate <60) as determined by history and/or serum basic metabolic panel
* Neurogenic detrusor hyperreflexia, detrusor areflexia, detrusor sphincter dyssynergia, chronic urinary catheterization

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Ambulatory Urogynecology Clinic
Sampling Method: Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2014-01; Primary Completion 2014-01 (Estimated)

PRIMARY OUTCOMES:
Impact of surgical treatment of apical pelvic organ prolapse on bothersome nocturia. | 1 year
  To evaluate whether women with bothersome pre-operative nocturia who undergo surgical treatment for their POP will demonstrate significant symptomatic improvement in nocturia as measured by the NNES-Q questionnaire.

SECONDARY OUTCOMES:
Impact of surgical treatment of apical pelvic organ prolapse on nocturnal polyuria. | 1 year
  To evaluate whether women with bothersome pre-operative nocturia who undergo surgical treatment for their POP will demonstrate a significant post-operative improvement in their nocturnal polyuria based on voiding diaries.
Impact of surgical treatment of apical pelvic organ prolapse on urine osmolality parameters. | 1 year
  To evaluate whether women with bothersome pre-operative nocturia who undergo surgical treatment for their POP will demonstrate a significant post-operative improvement in their ability to concentrate urine based on urine osmolality parameters.

CONTACTS AND LOCATIONS:
Overall Officials: Elizabeth Mueller, MD, Principal Investigator — Loyola University Medical Center Department of Urology and Obstetrics
Locations (1):
- Loyola University Medical Center, Maywood, Illinois, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Madersbacher S, Cornu JN. Nocturnal polyuria: it's all about definition, and be Patient! Eur Urol. 2013 Mar;63(3):548-50. doi: 10.1016/j.eururo.2012.10.043. Epub 2012 Nov 2. No abstract available. PMID 23141934
- [Background] Yanik FF, Akpolat T, Kocak I. Acute renal failure--an unusual consequence of uterine prolapse. Nephrol Dial Transplant. 1998 Oct;13(10):2648-50. doi: 10.1093/ndt/13.10.2648. No abstract available. PMID 9794579
- [Background] Gomes CM, Rovner ES, Banner MP, Ramchandani P, Wein AJ. Simultaneous upper and lower urinary tract obstruction associated with severe genital prolapse: diagnosis and evaluation with magnetic resonance imaging. Int Urogynecol J Pelvic Floor Dysfunct. 2001;12(2):144-6. doi: 10.1007/s001920170082. PMID 11374515
- [Background] Beverly CM, Walters MD, Weber AM, Piedmonte MR, Ballard LA. Prevalence of hydronephrosis in patients undergoing surgery for pelvic organ prolapse. Obstet Gynecol. 1997 Jul;90(1):37-41. doi: 10.1016/S0029-7844(97)00240-8. PMID 9207809
- [Background] Abbasy S, Kenton K. Obliterative procedures for pelvic organ prolapse. Clin Obstet Gynecol. 2010 Mar;53(1):86-98. doi: 10.1097/GRF.0b013e3181cd4252. PMID 20142646
- [Background] Bing MH, Moller LA, Jennum P, Mortensen S, Lose G. Validity and reliability of a questionnaire for evaluating nocturia, nocturnal enuresis and sleep-interruptions in an elderly population. Eur Urol. 2006 Apr;49(4):710-9. doi: 10.1016/j.eururo.2005.11.034. Epub 2006 Jan 13. PMID 16442700
- [Background] Chuang FR, Lee CH, Chen CS, Weng HH, Wang IK. Bilateral moderate hydroureteronephrosis due to uterine prolapse: two case reports and review of the literature. Ren Fail. 2003 Sep;25(5):879-84. doi: 10.1081/jdi-120024303. PMID 14575296
- [Background] Floyd MS Jr, Casey RG, Bredin HC. Procidentia: a reversible cause of hydronephrosis in an 80-year-old woman. Int Urogynecol J Pelvic Floor Dysfunct. 2008 Aug;19(8):1179-81. doi: 10.1007/s00192-008-0587-x. Epub 2008 Mar 11. PMID 18330482